CLINICAL TRIAL: NCT02039375
Title: Optimal Post Tpa-Iv Monitoring in Ischemic STroke
Brief Title: Safety Study of Post Intravenous tPA Monitoring in Ischemic Stroke
Acronym: OPTIMIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00087038
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Ischemic Stroke
Keywords: IV tPA; Thrombolysis; Stroke; Ischemic; Monitoring
MeSH Terms: conditions — Stroke; Ischemic Stroke; Ischemia

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- "Hopkins" post tPA monitoring protocol (Experimental): Patients treated with IV tPA (intravenous tissue Plasminogen Activator) for acute stroke will be monitored in a non-ICU setting following the "Hopkins" post tPA monitoring protocol, a new schedule for vital signs and neurochecks. These patients will have vital signs and neurochecks every 15 minutes for two hours, then once upon admission to the stroke unit and after one hour, then every two hours for 8 hours and then every four hours until 24 hours post tPA.
  Interventions: Other: "Hopkins" post tPA for ischemic stroke monitoring protocol

INTERVENTIONS:
Other: "Hopkins" post tPA for ischemic stroke monitoring protocol — The "Hopkins" post tPA monitoring protocol includes: vital signs and neurochecks, per standard of care for the first two hours (every 15 minutes), then on arrival to unit, in one hour, every 2 hours for 8 hours, and every 4 hours to complete 24 hours.

SUMMARY:
Intravenous (IV) tissue plasminogen activator (tPA) is the only FDA-approved therapy for treatment of acute ischemic stroke. In the United States, IV tPA is typically administered in the Emergency Department (ED) for patients presenting with acute ischemic stroke within 4.5 hours of symptom onset. It is current practice that post-tPA patients are monitored in an intensive care unit or intensive care unit (ICU)-like setting for at least 24 hours, in part due to frequent vital sign and neurological monitoring that is currently the standard of care. However, rigorous evidence to support this practice is largely lacking. In a retrospective analysis of 153 patients receiving IV tPA at Johns Hopkins Hospital (JHH) and Johns Hopkins Bayview Medical Center (JHBMC), investigators have shown that most patients who have ICU needs in the first 24 hours after tPA administration develop such needs by the end of the tPA infusion. Patients without ICU needs by the end of the tPA infusion, do not require further ICU resources if patients' presenting NIH Stroke Scale (NIHSS) is below 10. This study is a prospective clinical trial that aims at establishing the first proof-of-concept and feasibility of whether patients with a low NIHSS (NIHSS 9 or less) and that do not need ICU care by the end of the tPA infusion, can be monitored safely in a non-ICU setting with a novel monitoring protocol. Identifying post-tPA patients who can be safely monitored in a non-ICU environment may improve cost-effective utilization of ICU resources and reduce the length of hospitalization for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent (or a Legally Authorized Representative (LAR) available to provide informed consent) and comply with study assessments for the full duration of the study.
* Age 18-80 years
* Patients to be included will be diagnosed as having an acute ischemic stroke by history and physical exam and receive IV tPA within 4.5 hours of symptom onset according to current guidelines for acute stroke care.
* NIHSS at presentation <10
* Patients do not have ICU needs in the judgment of the treating ED physician or neurologist by the end of the tPA infusion
* NIHSS at the end of tPA infusion <10

Exclusion Criteria:

* For patients receiving IV tPA according to the current standard of care, the following exclusion criteria apply:

  * Age <17 or >80
  * ICU need or indication by the end of the tPA infusion
  * NIHSS >9 at presentation or at the end of the tPA infusion
  * Indication/need for endovascular recanalization therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor C Urrutia, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Faigle R, Sharrief A, Marsh EB, Llinas RH, Urrutia VC. Predictors of critical care needs after IV thrombolysis for acute ischemic stroke. PLoS One. 2014 Feb 12;9(2):e88652. doi: 10.1371/journal.pone.0088652. eCollection 2014. PMID 24533130
- [Result] Faigle R, Butler J, Carhuapoma JR, Johnson B, Zink EK, Shakes T, Rosenblum M, Saheed M, Urrutia VC. Safety Trial of Low-Intensity Monitoring After Thrombolysis: Optimal Post Tpa-Iv Monitoring in Ischemic STroke (OPTIMIST). Neurohospitalist. 2020 Jan;10(1):11-15. doi: 10.1177/1941874419845229. Epub 2019 May 5. PMID 31839859
- See also: Preliminary work — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0088652

RESULTS

PARTICIPANT FLOW:
Groups:
- "Hopkins" Post tPA Monitoring Protocol: Patients treated with IV tissue plasminogen activator (tPA) for acute stroke will be monitored in a non-ICU setting following the "Hopkins" post tPA monitoring protocol, a new schedule for vital signs and neurochecks. These patients will have vital signs and neurochecks every 15 minutes for two hours, then once upon admission to the stroke unit and after one hour, then every two hours for 8 hours and then every four hours until 24 hours post tPA.
  "Hopkins" post tPA for ischemic stroke monitoring protocol: The "Hopkins" post tPA monitoring protocol includes: vital signs and neurochecks, per standard of care for the first two hours (every 15 minutes), then on arrival to unit, in one hour, every 2 hours for 8 hours, and every 4 hours to complete 24 hours.
Period: Overall Study
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
Started | 35
Completed | 33
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- "Hopkins" Post tPA Monitoring Protocol: Patients treated with IV tPA for acute stroke will be monitored in a non-ICU setting following the "Hopkins" post tPA monitoring protocol, a new schedule for vital signs and neurochecks. These patients will have vital signs and neurochecks every 15 minutes for two hours, then once upon admission to the stroke unit and after one hour, then every two hours for 8 hours and then every four hours until 24 hours post tPA.
  "Hopkins" post tPA for ischemic stroke monitoring protocol: The "Hopkins" post tPA monitoring protocol includes: vital signs and neurochecks, per standard of care for the first two hours (every 15 minutes), then on arrival to unit, in one hour, every 2 hours for 8 hours, and every 4 hours to complete 24 hours.
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
Number analyzed (Participants) | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Needing ICU Care/Interventions Within the First 24 Hours of IV tPA Administration
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
Number analyzed (Participants) | 35
Participants | 0

2. Secondary Outcome: Severity of Stroke at 24 Hours as Assessed by the National Institutes of Health Stroke Scale (NIHSS)
Description: The NIHSS is a scale of stroke severity with 15 items and a score range from 0 to 42. 0 = no stroke; 1-4 = minor stroke; 5-15 = moderate stroke; 15-20 = moderate/severe stroke; 21-42 = severe stroke.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
Number analyzed (Participants) | 35
score on a scale | 1 [0 to 3]

3. Secondary Outcome: Degree of Disability as Assessed by the Modified Rankin Score (mRS)
Description: The mRS is a scale of disability with a score range from 0-6. 0 - no symptoms, back to normal.
  1. - some symptoms, able to do all prior activities, does not need help from others.
  2. - some symptoms, unable to do all prior activities, does not need help from others.
  3. - needs help from others, able to walk.
  4. - needs help from other, unable to walk without help.
  5. - needs total care.
  6. - the patient has expired.
Time Frame: At the time of discharge from the hospital, up to 90 days
Measure: Median (Full Range); unit: score on a scale
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
Number analyzed (Participants) | 35
score on a scale | 1 [0 to 3]

4. Secondary Outcome: Severity of Symptoms of Stroke at 90 Days as Assessed by the NIHSS
Description: as for outcome 2
Time Frame: At 90 days
Population: The NIHSS assessment at 90 days was not done for 7 participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
Number analyzed (Participants) | 28
score on a scale | 0 [0 to 1]

5. Secondary Outcome: Degree of Disability at 90 Days as Assessed by the mRS
Description: The mRS is a scale of disability with a score range from 0-6. 0-no symptoms, back to normal.
  1. some symptoms, able to do all prior activities, does not need help from others.
  2. some symptoms, unable to do all prior activities, does not need help from others.
  3. needs help from others, able to walk.
  4. needs help from other, unable to walk without help.
  5. needs total care.
  6. the patient has expired.
Time Frame: At 90 days
Measure: Median (Full Range); unit: score on a scale
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
Number analyzed (Participants) | 33
score on a scale | 0 [0 to 6]

6. Secondary Outcome: Mortality at 90 Days
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
Number analyzed (Participants) | 35
Participants | 1

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | "Hopkins" Post tPA Monitoring Protocol
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | "Hopkins" Post tPA Monitoring Protocol (N=35)
Mortality (Cardiac disorders) | 1 (1) — One patient died several weeks after discharge from a cardiovascular event unrelated to his stroke or the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT02039375/Prot_SAP_000.pdf